CLINICAL TRIAL: NCT02942901
Title: Clinical Evaluation of PET-CT for Staging of Colorectal Lung Metastases - a Prospective Monocentric Feasibility Study
Brief Title: Clinical Evaluation of PET-CT for Staging of Colorectal Lung Metastases
Status: Completed | Type: Observational
Sponsor: Lung Clinic Heckeshorn (Other)
Responsible Party: Sponsor
Other Study IDs: Oskar Helene 11/2016
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: PET-CT; pulmonary metstasectomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PET-CT

SUMMARY:
Surgery has been available for the treatment of pulmonary metastases in metastatic colorectal cancer and promising overall survival was observed in retrospective studies with selected patients. This study investigated whether the preoperative FDG- PET/CT scan influences survival in this patient group. Furthermore, we tried to identify other prognostic factors associated with overall survival and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with pulmonary metastases eligible for pulmonary metastasectomy

Exclusion Criteria:

* Second primary cancer within the last 2 years (exception basal cell carcinoma of the skin)
* Pregnancy,
* Drug addiction,
* Renal dialysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary metastases eligible for pulmonary metastasectomy
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Number and sites of metastases detected by PET-CT | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Lung Clinic Heckeshorn at HELIOS Hospital Emil von Behring, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pastorino U, Veronesi G, Landoni C, Leon M, Picchio M, Solli PG, Leo F, Spaggiari L, Pelosi G, Bellomi M, Fazio F. Fluorodeoxyglucose positron emission tomography improves preoperative staging of resectable lung metastasis. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1906-10. doi: 10.1016/s0022-5223(03)00211-3. PMID 14688704